CLINICAL TRIAL: NCT03686332
Title: PERICLES (PEnile Cancer Radio- and Immunotherapy CLinical Exploration Study)-a Phase 2 Study of Atezolizumab With or Without Radiotherapy in Penile Cancer
Brief Title: PEnile Cancer Radio- and Immunotherapy CLinical Exploration Study
Acronym: PERICLES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N18PER; 2018-000603-17 (EudraCT Number)
Record Dates: First submitted 2018-09-18; First posted 2018-09-26 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Penile Cancer
Keywords: Radiotherapy; Immunotherapy; Atezolizumab
MeSH Terms: conditions — Penile Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: All patients included will have unresectable advanced penile cancer. Patients will be discussed in multi-disciplinary rounds to establish this criterion. Two treatment groups will be distinguished.
  Arm A: Patients with locoregional lymph node disease who have not received extensive inguinal or pelvic irradiation on the involved area before. Patients in this group will concurrently be treated with locoregional radiotherapy and atezolizumab.
  Arm B: Patients who are not expected to derive benefit from radiotherapeutic treatment. This group will mainly consist of patients with distant metastases or previously treated locoregional disease and will only be treated with atezolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezolizumab and Radiotherapy (Other): Patients in this group will concurrently be treated with locoregional radiotherapy and atezolizumab.
  Drug: Arm A: Atezolizumab and Radiotherapy
  Atezolizumab, 1200 mg, every 3 weeks, by IV infusion and receive 33 fractions of 1.5 or 1.8 Gy irradiation.
  Interventions: Drug: Arm A: Atezolizumab and Radiotherapy; Drug: Arm B: Atezolizumab
- Arm B: Atezolizumab (Other): Atezolizumab, 1200 mg, every 3 weeks, by IV infusion.
  Interventions: Drug: Arm A: Atezolizumab and Radiotherapy; Drug: Arm B: Atezolizumab

INTERVENTIONS:
Drug: Arm A: Atezolizumab and Radiotherapy — patients will receive atezolizumab, 1200 mg, every 3 weeks, by IV infusion. Patients in group A will additionally receive 33 fractions of 1.5 (locoregional affected lymph nodes) and 1.8 Gy (tumor+margin) irradiation, concurrently with atezolizumab treatment.
Drug: Arm B: Atezolizumab — patients will receive atezolizumab, 1200 mg, every 3 weeks, by IV infusion.

SUMMARY:
Patients with advanced penile cancer have a poor prognosis (21% 2-year overall survival from moment of diagnosis) and high morbidity due to progressive locoregional disease.

Translational studies show high rates of infiltrating immune cells and PD-L1 positivity, suggesting that immunotherapy may be beneficial in this disease. Atezolizumab, targeting PD-L1, is active in several cancer types and is generally well-tolerated. This study will investigate whether atezolizumab can be combined with radiotherapy to control locoregional lymph node disease. Furthermore, the activity of atezolizumab in advanced penile cancer patients will be investigated.

DETAILED DESCRIPTION:
Rationale Patients with advanced penile cancer have a poor prognosis (21% 2-year overall survival from moment of diagnosis) and high morbidity due to progressive locoregional disease.

Translational studies show high rates of infiltrating immune cells and PD-L1 positivity, suggesting that immunotherapy may be beneficial in this disease. Atezolizumab, targeting PD-L1, is active in several cancer types and is generally well-tolerated. This study will investigate whether atezolizumab can be combined with radiotherapy to control locoregional lymph node disease. Furthermore, the activity of atezolizumab in advanced penile cancer patients will be investigated.

Objectives:

1. Efficacy of atezolizumab in advanced penile cancer patients.
2. Feasibility of a protracted schedule of radiotherapy on locoregional disease in combination with immunotherapy for advanced penile cancer

Study design:

Single-center, nonrandomized, Phase 2 study with 2 treatment arms.

Study population:

Men, ≥18 years of age, with advanced inoperable penile cancer, N=32.

Intervention:

All patients will receive atezolizumab, 1200 mg, every 3 weeks, by IV infusion. Patients in group A will additionally receive 33 fractions of 1.5 (locoregional affected lymph nodes) and 1.8 Gy (tumor+margin) irradiation, concurrently with atezolizumab treatment.

Primary endpoint:

Progression-free survival at 1 year.

Main secondary endpoint:

2-year overall survival rate of the complete study population. Percentage of patients who complete the full course of radiotherapy in the radiotherapy/atezolizumab arm.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will be treated every 3 weeks with atezolizumab for one year or until loss of clinical benefit. Atezolizumab is generally well tolerated although immune-related toxicity does occur.

Toxicity of combining atezolizumab with a long course of radiotherapy is unknown and may result in increased toxicity. It is unknown whether atezolizumab will induce responses in patients with advanced penile cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, prior to performing any protocol-related procedures, including screening evaluations.
* Age > 18 years at time of study entry.
* Advanced histologically documented, squamous cell carcinoma of the penis or distal urethra. Advanced disease is defined as:
* Distant metastases, OR
* LRAPC, defined as a large or inoperable primary tumor (T4), palpable nodes >3cm in diameter or fixed nodes, suspicion of extra-nodal extension or pelvic node involvement (N2/N3)
* Arm A: Locoregional disease (with or without distant metastases), likely to derive benefit from locoregional radiotherapy and not previously treated with radiotherapy.
* Arm B: Benefit of locoregional radiotherapy unlikely OR previously treated with irradiation.
* World Health Organisation (WHO) performance status of 0 or 1.
* Life expectancy of > 12 weeks.
* Adequate normal organ and marrow function as defined below:
* Haemoglobin ≥ 5.6/mmol/L
* White blood cell count (WBC) ≥ 2 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L (>100,000 per mm3)
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome, who will be allowed in consultation with a study physician.
* AST/ALT ≤ 2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤ 5x ULN.
* Serum creatinine clearance >30 mL/min by calculation with the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection measurement.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both Roche staff and/or staff at the study site) or previous enrolment in the present study.
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a PD-1 or PD-L1 inhibitor
* History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of study drug
* Low potential risk of 3-year cancer-specific death (estimated<5%), including adequately treated non-melanoma skin cancer without evidence of disease, adequately treated carcinoma in situ without evidence of disease, or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 7 and PSA < 10 ng/mL) undergoing active surveillance.
* Treatment with the last dose of any systemic anti-cancer therapy ≤ 21 days prior to the first dose of study drug. Local treatment of isolated lesions for palliative intent is acceptable (eg, local surgery or radiotherapy).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at doses ≤10 mg/day of prednisone, or an equivalent corticosteroid.
* History of primary immunodeficiency, allogeneic organ transplant or autoimmune disease, including - but not limited to - myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone will not be excluded from this study. Patients with controlled diabetes mellitus type I on a stable dose of insulin regimen may be eligible for this study.
* Uncontrolled significant intercurrent illness, including - but not limited to - ongoing or active infection (including acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV)), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known active tuberculosis
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Brain metastases or leptomeningeal disease. Inclusion of patients with brain metastases is allowed if patients have been adequately treated, are not symptomatic and show no signs of progression on brain imaging 28 days after completion of treatment (including surgery, radiotherapy or treatment with systemic corticosteroids).
* Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 1 year. | 1 year
  Progression-free survival at 1 year.

SECONDARY OUTCOMES:
2-year overall survival rate of the complete study population. | 2 year
  The key secondary outcome measure will be 2-year overall survival rate in the full study cohort (Arm A and B combined).
  radiotherapy/atezolizumab arm.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel MS van der Heijden, Dr., Principal Investigator — NKI-AvL
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] de Vries HM, Rafael TS, Gil-Jimenez A, de Feijter JM, Bekers E, van der Laan E, Lopez-Yurda M, Hooijberg E, Broeks A, Peters D, Seignette IM, Pos FJ, Horenblas S, van Rhijn BWG, Jordanova ES, Brouwer OR, Schaake E, van der Heijden MS. Atezolizumab With or Without Radiotherapy for Advanced Squamous Cell Carcinoma of the Penis (The PERICLES Study): A Phase II Trial. J Clin Oncol. 2023 Nov 1;41(31):4872-4880. doi: 10.1200/JCO.22.02894. Epub 2023 Jul 24. PMID 37487169